CLINICAL TRIAL: NCT03516747
Title: Ultrasound Guided Fine Needle Aspiration of Parathyroid Gland as a Pre Operative Localization Tool to Identify Pathological Parathyroid
Brief Title: Preoperational Fine Needle Aspiration of Pathological Parathyroid Gland
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: we gave up
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, Paker Miki, Dr.paker miki. principal investigator, HaEmek Medical Center, Israel
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 18-0005-EMC
Record Dates: First submitted 2018-04-03; First posted 2018-05-04 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: Parathyroid Adenoma; Hypercalcemia
Keywords: cytology; parathyroidectomy; parathyroid hormone level
MeSH Terms: conditions — Parathyroid Neoplasms; Hypercalcemia

STUDY DESIGN:
Intervention Model Description: open label, non- randomised, prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- investigation group (Experimental): participants that suffer hypercalcemia due to primary hyperparathyroidism. include all participants in the trial
  Interventions: Diagnostic Test: pre operative parathyroid hormone level measurement; Diagnostic Test: pre operative parathyroid cytology; Diagnostic Test: parathyroid hormone level measurement; Diagnostic Test: parathyroid cytology

INTERVENTIONS:
Diagnostic Test: pre operative parathyroid hormone level measurement — At the clinic, the participants will undergo ultrasound examination with fine needle aspiration. The aspirated material will be sent for parathyroid hormone level measurement.
Diagnostic Test: pre operative parathyroid cytology — At the clinic, the participants will undergo neck ultrasound examination with fine needle aspiration. The aspirated material will be sent for cytology examination.
Diagnostic Test: parathyroid hormone level measurement — At surgery, after the pathologic gland is excised , the gland will be aspirated. The material will be sent for parathyroid hormone level measurement.
Diagnostic Test: parathyroid cytology — At surgery, after the pathologic gland is excised , it will be aspirated again for cytologic examination.

SUMMARY:
Identification and localization of pathological parathyroid gland before parathyroidectomy is traditionally done by a combination of two methods: ultrasound and sestamibi scan. The investigators would like to show that one exam that includes ultrasound and fine needle aspiration of the parathyroid gland for parathyroid hormone level is as accurate as the traditional method.

DETAILED DESCRIPTION:
A prospective, open label, single arm trial that includes participants that suffer hypercalcemia due to primary hyperparathyroidism and are candidates for parathyroidectomy.

participants visit the investigator's head and neck clinic. the investigator confirms that the participant has an indication for parathyroidectomy according to the official criteria. Later on, the investigator looks at the localization tests that have already been done (neck ultrasound and MIBI [methoxyisobutyllisonitrile] scan) in order to plan the surgery. In case participant has not made those tests- the investigator fills a written request to do so. then, the investigator will perform a neck ultrasound and identifies the pathological parathyroid gland. The suspected pathological gland is aspirated using a 27 gauge needle attached to a 5 cc syringe fills with 1 cc saline (0.9% NaCL) under the guidance of the ultrasound. The aspirated material is sent for 2 examinations:

1. parathyroid hormone level: the aspirated material is injected into a ethylenediaminetetraacetic acid (EDTA) vial and send to the hospital's endocrine laboratory. the parathyroid hormone level is processed using chemiluminescence method and represented in Pg/ml units.
2. cytology examination. The aspirated material is spread on a glassed slide and prepared with a Giemsa stain for a cytologic examination. cytologic features such as cell type, cytoplasmic characteristics,cell block structure and chromatin appearance is addressed by the pathologist.

After completion of the ultrasound - guided needle aspiration the participant is given an exact date for the surgery.

The surgery is carried out routinely with the same surgical steps that the investigator is familiar with. At the end of surgery, after the pathological parathyroid gland was extracted from the neck, it is aspirated with a 27Gy needle attached to a 5 cc, syringe filled with a 1 cc saline (0.9% NaCL).

The aspirated material is sent to the same, above mentioned, examinations (parathyroid hormone level and cytology).

After the investigator receives the final pathological result of the suspected gland and confirm that the excised tissue was indeed a pathological parathyroid one, the investigators are able to answer 2 important questions:

1. Is high level of parathyroid hormone which was aspirated from a suspected pathological parathyroid tissue is a good indicator that the tissue is indeed a pathological parathyroid.
2. Is there a difference between parathyroid cytology of a tissue aspirated transcutaneously to a parathyroid cytology of material aspirated directly from the parathyroid gland.

ELIGIBILITY:
Inclusion Criteria:

* above 18 years old
* participants that suffer from primary hyperparathyroidism with an indication for parathyroidectomy

Exclusion Criteria:

* Chronic renal failure
* kidney transplant participant
* MEN (multiple endocrine neoplasia) syndrome
* pregnancy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-06-09 (Actual); Primary Completion 2020-04-09 (Actual); Study Completion 2020-08-09 (Actual)

PRIMARY OUTCOMES:
parathyroid hormone level from a pathological parathyroid gland | one month after the patient starts the study
  Under ultrasound guidance, the investigators will locate a neck leison which based on previous localization imaging modalities, is proven to be a pathological parathyroid gland.The investigators will aspirate material from this gland and send it for measurement of parathyroid hormone level. we will prove that a lesion that contains high levels of parathyroid hormone is indeed a parathyroid gland. thereby, this method may replace other localization methods
parathyroid hormone level from a pathological parathyroid gland | one month after the patient starts the study
  At surgical final step, after the pathological parathyroid gland is ex vivo the investigator will aspirate material from it and send it for measurement of parathyroid hormone level. we will prove that a lesion that contains high levels of parathyroid hormone is indeed a parathyroid gland.

SECONDARY OUTCOMES:
parathyroid gland cytology from a pathological parathyroid gland. | one month after the patient starts the study
  Under ultrasound guidance, the investigators will locate a neck leison which based on previous localization imaging modalities, is proven to be a pathological parathyroid gland.The investigators will aspirate material from this gland and send it for cytology examination.By doing so we will investigate whether cytology that was aspirated from parathyroid gland trans cutaneously is different from a cytology of the gland aspirated directly (ex vivo-after it the gland excised from the body).
parathyroid gland cytology | one month after the patient starts the study
  At surgical final step, after the pathological parathyroid gland is ex vivo the investigator will aspirate material from it and send it for cytology examination.By doing so the investigators will determine whether cytology that was aspirated from parathyroid gland trans cutaneously is different from a cytology of the gland aspirated directly (ex vivo- after it the gland excised from the body).

CONTACTS AND LOCATIONS:
Overall Officials: Dror Ashkenazi, M.D, Study Director — haemek medical center
Locations (1):
- Haemek Medical Center, Afula, Israel

IPD SHARING:
Plan to Share IPD: No
The investigators will not make individual participant data available due to the desire to preserve the privacy of the participants in the study